CLINICAL TRIAL: NCT00210886
Title: A Multicenter, Double-blind, Randomized Study to Compare the Efficacy and Safety of Levofloxacin 750 mg Once Daily for Five Days Versus Ciprofloxacin Twice Daily for Ten Days in the Treatment of Complicated Urinary Tract Infection and Acute Pyelonephritis.
Brief Title: A Comparison of the Effectiveness and Safety of Levofloxacin to That of Ciprofloxacin in Treating Complicated Urinary Tract Infection and Acute Pyelonephritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004705
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Tract Infections; Pyelonephritis
Keywords: complicated urinary tract infection; urinary tract infection; acute pyelonephritis; pyelonephritis; kidney infection; bladder infection
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis; Cystitis | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of two antibiotics in the treatment of complicated urinary tract infection or acute pyelonephritis (kidney infection). A 5-day course of 750 milligrams of levofloxacin given intravenously and/or by mouth once daily will be compared to a 10-day course of 400 milligrams of ciprofloxacin given intravenously and/or 500 milligrams of ciprofloxacin given by mouth twice daily.

DETAILED DESCRIPTION:
Levofloxacin has been approved in both its oral and intravenous forms to treat a large number of infections caused by bacteria. Levofloxacin and other members of a class of antibiotics known as fluoroquinolones have been used successfully to treat urinary and kidney infections. This study will compare the effectiveness and safety of levofloxacin given for 5 days to that of another fluoroquinolone, ciprofloxacin, given for 10 days in treating complicated urinary tract infection or acute pyelonephritis (kidney infection). A shorter course of antibiotics may help patients take all of their medication, which is critically important for curing the infection. A shorter course may also help prevent the development of bacteria that cannot be killed by antibiotics. Patients will take 750 milligrams of levofloxacin intravenously and/or by mouth once daily for 5 days or 400 milligrams of ciprofloxacin intravenously and/or 500 milligrams of ciprofloxacin by mouth twice daily for 10 days. To prevent the study doctor, study staff and patients from knowing which study drug they are taking, all study drug will manufactured to look the same and patients on the 5-day regimen will be given placebo for the last 5 days of their participation in the study. The intravenous infusion bags will be covered so that the solution cannot be seen. The objective of the study is to demonstrate that 5 days of levofloxacin once daily is at least as effective as 10 days of ciprofloxacin twice daily in treating complicated urinary tract infection or acute pyelonephritis. Patients will take 750 milligrams of levofloxacin intravenously and/or by mouth once daily for 5 days or 400 milligrams of ciprofloxacin intravenously and/or 500 milligrams of ciprofloxacin by mouth twice daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Positive dipstick test for leukocyte esterase AND/OR at least 5 white blood cells per centrifuged urine sediment AND/OR at least 10 white blood cells per microliter of uncentrifuged urine
* outpatient or inpatient (in hospital, nursing home, or other extended-care facility)
* clinical diagnosis of either complicated urinary tract infection or acute pyelonephritis.

Exclusion Criteria:

* Allergy or serious adverse reaction to levofloxacin, ciprofloxacin, or other fluoroquinolone
* urinary tract surgery or lithotripsy (treatment for kidney stones) within 7 days before study entry
* a second coexisting bacterial infection that requires systemic antibiotics
* need for a second antibiotic to treat the urinary tract infection
* obstruction of the urinary tract
* prostate infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1109 (Actual)
Dates: Start 2004-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Combination of clinical success and microbiologic eradication (known as therapeutic response) at post-therapy visit.

SECONDARY OUTCOMES:
By patient and pathogen microbiologic and clinical responses at the post-therapy and post-study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Peterson J, Kaul S, Khashab M, Fisher AC, Kahn JB. A double-blind, randomized comparison of levofloxacin 750 mg once-daily for five days with ciprofloxacin 400/500 mg twice-daily for 10 days for the treatment of complicated urinary tract infections and acute pyelonephritis. Urology. 2008 Jan;71(1):17-22. doi: 10.1016/j.urology.2007.09.002. PMID 18242357
- [Result] Klausner HA, Brown P, Peterson J, Kaul S, Khashab M, Fisher AC, Kahn JB. A trial of levofloxacin 750 mg once daily for 5 days versus ciprofloxacin 400 mg and/or 500 mg twice daily for 10 days in the treatment of acute pyelonephritis. Curr Med Res Opin. 2007 Nov;23(11):2637-45. doi: 10.1185/030079907x233340. PMID 17880755
- [Result] Peterson J, Kaul S, Khashab M, Fisher A, Kahn JB. Identification and pretherapy susceptibility of pathogens in patients with complicated urinary tract infection or acute pyelonephritis enrolled in a clinical study in the United States from November 2004 through April 2006. Clin Ther. 2007 Oct;29(10):2215-21. doi: 10.1016/j.clinthera.2007.10.008. PMID 18042477
- [Derived] Mospan GA, Wargo KA. 5-Day versus 10-Day Course of Fluoroquinolones in Outpatient Males with a Urinary Tract Infection (UTI). J Am Board Fam Med. 2016 Nov 12;29(6):654-662. doi: 10.3122/jabfm.2016.06.160065. PMID 28076247
- See also: Levofloxacin Versus Ciprofloxacin in the Treatment of Complicated Urinary Tract Infection or Acute Pyelonephritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=626&filename=CR004705_CSR.pdf